CLINICAL TRIAL: NCT02614677
Title: To Advance the New Disability Evaluation System in Taiwan
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Clinical Professor, Changhua Christian Hospital
Other Study IDs: CCH-140713
Record Dates: First submitted 2015-11-08; First posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Motor Dysfunction
Keywords: Disability Evaluation System; SF-12; ICF model
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Before 2007, the disability evaluation was based on the medical model in Taiwan. According to the People with Disabilities Rights Protection Act announced on 11 July 2007, the assessment of a person's eligibility for disability benefits has to be determined as suffering one of eight malfunction categories based on the International Classification of Functioning, Disability, and Health (ICF) framework. People with disabilities want to issue a disability identification and other welfare & services need processes of evaluation & assessment based on the ICF framework for the evaluation report and result of living need by the committee composed of professionals from medicine, social work, special education and employment counseling and evaluation.

In this year, investigators planed the project with the Taiwan Society of ICF to develop the evaluation form. The experts from various disciplines of the ICF Office convened internal integration meetings to reach a consensus for developed the ICF evaluation form, add the code of pain and sleep and the items from Short-Form 12 for quality of life to the questionnaire. The results were used to analysis other relevant factors affecting the disability evaluation. And then add the core set from World Health Organization to both physical and mental disorders linked coding group, compared the new disability evaluation system and evaluate the living need of people with disability to provide suggestion for core set.

ELIGIBILITY:
Inclusion Criteria:

* comply with a standard of the disability evaluation

Exclusion Criteria:

* no

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with disabilities want to issue a disability identification
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assessment of Quality of life by disability evaluate system | One day when patients came first
Pain intensity on the Numerical Rating Scale | One day when patients came first

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Dawan, Changhua, Taiwan